CLINICAL TRIAL: NCT02777112
Title: The Effects of E-mental Health Program and Job Coaching on the Risk of Major Depression and Productivity in Canadian Male Workers
Brief Title: The Effects of E-mental Health Program and Job Coaching on the Risk of Major Depression in Canadian Working Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Movember Foundation (Other)
Responsible Party: Principal Investigator, JianLi Wang, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: #UCAL_01
Record Dates: First submitted 2016-05-11; First posted 2016-05-19 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Depression; Men
Keywords: high-risk; early prevention; productivity; return on investment; workplace; e-mental health program; job coach
MeSH Terms: conditions — Depression; Multiple Endocrine Neoplasia Type 1 | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Placebo Comparator): This group will receive generic information about depression and serve as control
  Interventions: Other: No intervention
- e-mental health program (Experimental): This group will receive the developed e-mental health program
  Interventions: Other: e-mental health program
- e-mental health program and job coaching (Experimental): This group will receive the developed e-mental health program plus interactive job coaching through telephone.
  Interventions: Other: e-mental health program and job coaching

INTERVENTIONS:
Other: e-mental health program — This program is delivered over the Internet, which includes modules of Information (about depression, workplace factors and alcohol use), Practical Tips (Cognitive Behavioral Therapy, Mindfulness relaxation, workplace strategies), Tools (for monitoring and predicting depression and occupational functioning), and Goal Setting and Tracking.
  Arms: e-mental health program
Other: e-mental health program and job coaching — This combines the e-mental health program and interactive job coaching delivered through telephone. The e-mental health program is delivered over the Internet, which includes modules of Information (about depression, workplace factors and alcohol use), Practical Tips (Cognitive Behavioral Therapy, Mindfulness relaxation, workplace strategies), Tools (for monitoring and predicting depression and occupational functioning), and Goal Setting and Tracking. The job coaching can be accessed by appointment.
  Arms: e-mental health program and job coaching
Other: No intervention — Receiving generic information about men's depression from the Movember Foundation website: https://ca.movember.com/programs/mental-health
  Other Names: control group
  Arms: Control

SUMMARY:
There is a pressing need for innovation in prevention of major depression in male workers. Major depression (MDE) affects workers' health and productivity. In the United States, workers with depression cost an estimated US $44.01 billion per year in lost productivity. One of the severe consequences of having MDE is potential suicide and Canadian national data showed that 76% of all suicides in 2009 were male. In the workplace, risk factors for having MDE differ for men and women. For instance, job strain, family to work conflict and job insecurity seem to be more prominent MDE risk factors in men than in women. Compounding men's risk, men are less likely than women to seek help and to disclose depressive symptoms and often delay help seeking until symptoms become severe. Men are socialized to be emotionally stoic and exemplify traditional masculine characteristics such as independence, self-reliance and dominance. Men are concerned over the perceived negative judgments from family and friends if they access treatment for depression. These gender specific experiences along with a limited knowledge base about effective interventions call for innovative solutions tailored for men. The proposed study was to evaluate the effectiveness of an e-mental health program on reducing the risk of major depression in Canadian working men.

DETAILED DESCRIPTION:
Primary Objective:

Among Canadian male workers who are at high risk of having major depressive episode (MDE), to evaluate the impacts of an e-mental health intervention and telephone-based job coaching on the 12-month risk proportion of MDE. MDE will be measured by the WHO's CIDI-SFMD.

Hypothesis: The risk proportions of MDE in the intervention groups will be lower than that in the control group over 12 months.

Secondary Objectives:

Among Canadian male workers who are at high risk of having MDE,

1. to evaluate the impacts of an e-mental health intervention and telephone-based job coaching on:

   * Changes in depression score
   * Changes in anxiety score
   * Changes in absenteeism
   * Changes in presenteeism
   * Return on investment
   * Predicted MDE risk

   Depression and anxiety scores will be measured by the Patient Health Questionnaire (PHQ-9) and the Generalized Anxiety Disorder (GAD-7), respectively. Absenteeism and presenteeism will be measured by the WHO's Health and Work Performance Questionnaire (HPQ).

   Hypothesis I: The reductions in depressive and anxiety scores in the intervention groups will be greater than those in the control group over 12 months.

   Hypothesis II: The means of negative changes in absenteeism and presenteeism scores in the intervention groups will be lower than those in the control group.

   Hypothesis III: Participants in the intervention groups will have greater reduction in predicted MDE risk than those in the control group.
2. To compare participants who receive e-mental health program only and those who receive e-mental health program and job coaching services in

   * One-year proportion of MDE
   * Changes in depression score
   * Changes in anxiety score
   * Changes in absenteeism
   * Changes in presenteeism
   * Return on investment
   * Predicted MDE risk

Hypothesis IV: The risk proportion of MDE in the e-mental health plus job coaching group will be lower than that in the e-mental health only group.

Hypothesis V: The reduction in depression and anxiety scores in the e-mental health plus job coaching group will be greater than those in the e-mental health program only group.

Hypothesis VI: The means of negative changes in absenteeism and presenteeism scores in the e-mental health plus job coaching group will be lower than those in the e-mental health program only group.

Hypothesis VII: Participants in the e-mental health plus job coaching group will have greater reduction in predicted MDE risk than those in the e-mental health program only group.

The proposed mixed-methods study is a prospective, intention-to-treat, randomized controlled trial with 3 arms:

* Control group (n = 400): individuals will receive general information about men's mental health
* Intervention arm 1 (n = 400): individuals will receive the e-mental health program.
* Intervention arm 2 (n = 400): individuals will receive the e-mental health program, and telephone based interactive work-life coaching.

An embedded qualitative interview component will be conducted with a sub sample of participants from the intervention groups to obtain in-depth perspectives about the effectiveness of interventions at the 12-month.

Recruitment and Screening will be contracted to a telephone interview firm that has access to the numbers of household landlines and cell phones across the country. Recruitment will be conducted using the method of Random Digit Dialing (RDD).

Online assessment: To ensure the use of the Internet, participants who complete the baseline telephone assessment are instructed to complete an online survey as the last step of the baseline assessment and informed consent. The online survey will include:

* A brief description of the purpose of the trial and commitment of privacy protection
* The Internet use (2 questions)
* The 12-item Job Content Questionnaire used in the Statistics Canada survey to measure self-reported work stress
* Consent and submission.

Randomization. Participants who complete the baseline telephone and online surveys will be randomized into intervention and control groups. The randomization will be conducted and managed by the project coordinator affiliated with the project.

1200 random numbers (between 0 and 1) will first be generated using Excel ("RAND()") for 1200 study identification numbers (ID), ranging from 1 to 1200. The 1200 random numbers will then be sorted at the descending order and categorized into 3 equal groups:

* the ID numbers in the first group (n = 400) will be allocated to the control group
* the ID numbers in the second group (n = 400) will be allocated to the e-mental health program only
* the ID numbers in the third group (n = 400) will be allocated to the e-mental health group plus job coaching.

The Excel sheet with ID numbers and random numbers will be kept and printed out for randomization.

For example, a participant is the 3rd one who completes the online survey, which is determined by the date of completion. The project coordinator will search for ID #3 on the Excel sheet. The ID #3 is in the second group. This participant will be assigned to the group that will receive e-mental health program only.

The date of randomization will be documented. Any outcomes/changes that occur after the randomization will be counted to the groups, regardless of course of the e-mental health and job coaching interventions and if the interventions are used by the participants.

After randomization, the project coordinator will contact the participant by email. For those in the control group, the email will include a link to the men's mental health page of the Movember Foundation website; for those in the e-mental health only group, the email will include a link to the e-mental health program log-in page, and the user name. Password will be send in a separate email; for those in the e-mental health plus job coaching group, the email will include a link to the page for e-mental health program and appointment booking system, and the user name. Password will be send in a separate email.

After randomization, a package including the following materials will be mailed to the participants:

* A thank-you letter
* the Movember Foundation web site link to men's mental health: https://ca.movember.com/mens-health/mental-health
* $20 incentive as appreciation of their participation.

The project coordinator will not be involved in follow-up data collection.

Follow-up assessments: The post-randomization assessments will be conducted at 6 months and 12 months by interviewers at the Mathison Centre for Mental Health & Education, University of Calgary.

To obtain in-depth information about how the e-mental health solution affects men's behaviors and risk profile, qualitative interviews will be conducted via telephone with 10% of participants in the intervention groups at the end of the randomized controlled trial (RCT) (i.e., after the 12-month assessment). The participants will represent those with diverse outcomes (clinical and occupational trajectories, and employment status changes). Qualitative interview data will yield in-depth data about the impacts of receiving the e-mental health solution and depression risk information on the outcomes. These data will be used to support and interpret the primary quantitative data base. The multiple forms of evidence generated through mixed methods designs are particularly useful for illuminating complex health issues.36

Data management: The telephone interview firm will transfer password protected baseline data to the PI on a monthly basis. The group assignment data will be transferred in a separate file. The 6- and 12-month follow-up assessments will be conducted at the telephone interview laboratory at the Mathison Centre for Mental Health Research & Education (the Centre), University of Calgary. There are 5 trained telephone interviewers. Of whom, 2 can conduct interviews in English and French. The laboratory has 5 stations which are equipped with the Computer Assisted Telephone Interview provided by the VOXCO company. One month before the scheduled follow-up interviews, letters will be sent to the participants to remind them of the upcoming interview. An interview log will be developed for each participant to document interview time, schedule, call-back, contact information and for the interviewer to make comments.

Over the course of the trial, the principal investigator (PI) and research staff will examine the data on a regular basis by running cross tabulation, frequency distribution and estimation of means and proportions to ensure the quality of the data and identify missing values and potential outliers. If missing values and outliers are found, the records will be referred back to the interviewer for clarification or call-back.

After the 12-month interview, participants' group status will be linked with interview data by study identification (ID) numbers. Over the study period, the investigators and the interviewers who conduct the follow-up interviews in Calgary will not have access to participants' group status. The interviewers who conduct the baseline assessment and randomization, will not be involved in follow-up interviews.

The PI and project coordinator will be responsible for maintaining the data and data quality control. A sub-committee has been formed for this trial. The committee members will communicate via teleconference at bi-monthly basis to review and discuss the progress, operational issues, data analysis and preliminary results.

ELIGIBILITY:
Inclusion Criteria:

* At the time of recruitment, working for pay
* At the time of recruitment and baseline assessment, have a high risk of having major depressive episode (MDE) based on our prediction algorithm. For the proposed study, 6.51+% will be defined as high risk for men
* May have MDE in the past 12 months, but in remission for at least 2 months prior to the study
* Have no language barriers to English or French
* Have access to the internet
* Provide email and mailing address

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1133 (Actual)
Dates: Start 2016-09; Primary Completion 2018-10 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Risk proportion of major depressive episode (MDE) over 12 months | 12-month follow-up assessment
  MDE occurred over the 12-month follow-up period will be measured by the Composite International Diagnostic Interview

SECONDARY OUTCOMES:
Change in depression score | 6- and 12-month follow-up assessment
  Depression score will be measured by the Patient Health Questionnaire (PHQ-9)
Change in presenteeism | baseline, 6- and 12-month follow-up assessment
  To be measured by the World Health Organization (WHO)'s Health and Work Performance Questionnaire
Change in absenteeism | baseline, 6- and 12-month follow-up assessment
  To be measured by the WHO's Health and Work Performance Questionnaire
Return on investment | baseline, 6- and 12-month follow-up assessment
  To be measured by the WHO's Health and Work Performance Questionnaire
Change in anxiety score | baseline, 6- and 12-month follow-up assessment
  Anxiety score will be measured by the Generalized Anxiety Disorder - 7 (GAD-7)

OTHER OUTCOMES:
Change in sleep disturbance | baseline, 6- and 12-month follow-up assessment
  To be measured by the scale of the PROMIS
Change in anger | baseline, 6- and 12-month follow-up assessment
  To be measured by the scale of the PROMIS

CONTACTS AND LOCATIONS:
Overall Officials: JianLi Wang, Principal Investigator — University of Calgary
Locations (1):
- Mathison Centre for Mental Health Research and Education, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Need to discuss with the ethics review board regarding the format of data sharing.

REFERENCES:
- [Derived] Wang J, Patten SB, Lam RW, Attridge M, Ho K, Schmitz N, Marchand A, Lashewicz BM. The Effects of an E-Mental Health Program and Job Coaching on the Risk of Major Depression and Productivity in Canadian Male Workers: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2016 Nov 15;5(4):e218. doi: 10.2196/resprot.6350. PMID 27847352